CLINICAL TRIAL: NCT05613868
Title: A Phase 2a Study of TPN-101 in Patients With Aicardi-Goutières Syndrome (AGS)
Brief Title: TPN-101 in Aicardi-Goutières Syndrome (AGS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Transposon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPN-101-AGS-201
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Aicardi-Goutières Syndrome (AGS)
Keywords: AGS; TPN-101; censavudine

STUDY DESIGN:
Intervention Model Description: open label, single group
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active, TPN-101 (Experimental): 100 mg/day to 400mg/ study investigational drug TPN-101 once daily for 48 weeks followed by 12 weeks of follow-up period.
  Interventions: Drug: TPN-101

INTERVENTIONS:
Drug: TPN-101 — 100 mg/ day up to 400mg/day of TPN-101
  Other Names: censavudine

SUMMARY:
A phase 2a multi-center, open-label single dose level study of TPN-101 in Patients with Aicardi-Goutières Syndrome (AGS)

DETAILED DESCRIPTION:
The study is planned in pediatric and adult patients with AGS that are greater than 1 year and weigh at least 10 kg. The TPN-101 dose will be adjusted from 100 mg to 400 mg based on weight to achieve similar drug exposures in all subjects. The study plans to enroll 10 - 16 subjects. This study includes a 6-8 week Screening Period, a 48-week Open label Treatment Period, and a 12-week Follow-up Period.

ELIGIBILITY:
Patients must meet all of the following criteria:

Inclusion

1. Male or female participants of the following ages:

   1. Cohort 1: Adults (≥ 18 years of age)
   2. Cohort 2: Adolescents (12 to 17 years of age)
   3. Cohort 3: Children 5 to 11 years of age
   4. Cohort 4: Children 1 to < 5 years of age and >= 10 kg in weight
2. Molecular diagnosis of AGS due to biallelic mutations in 1 of the following 5 genes: TREX1, RNASEH2A, RNASEH2B, RNASEH2C, or SAMHD1, or due to a recognized dominant mutation in TREX1
3. IFN score in peripheral blood > 2 standard deviations above the mean score of healthy controls measured on 3 occasions, approximately 2 weeks apart, during the 6-week Screening Period.
4. Clinical syndrome consistent with AGS diagnosis based on clinical, CSF, and radiological findings. The following are examples of such findings (none of these are required for inclusion):

   1. Early onset encephalopathy with psychomotor delay, spasticity, extrapyramidal signs, and microcephaly, the latter appearing in the first year of life
   2. Calcifications particularly visible at basal ganglia level (putamen, pallidus, and thalamus), but also extending to the periventricular white matter
   3. Cerebral white matter abnormalities
   4. Cerebral atrophy
   5. Important systemic symptoms in the early stages of the disease including irritability, feeding and sleeping difficulties, unexplained fevers, and the appearance of chilblain-like skin lesions on the fingers, toes, and ears
5. Has a reliable caregiver to accompany the patient to all study visits. Caregiver must have frequent contact with patient and be willing to monitor the patient's health and concomitant medications throughout the study

Exclusion Criteria:

1. Mutation in IFIH1, ADAR1, LSM11, or RNU7-1.
2. Pre-/perinatal infections, in particular the TORCH complex (toxoplasmosis, rubella, cytomegalovirus, herpes simplex virus)
3. Presence of other significant neurological disorders; brain tumor or other space-occupying lesion; history of severe head injury
4. Clinically significant intercurrent illness, medical condition, physical or laboratory abnormality
5. Autoimmune disease requiring treatment or management (quiescent rheumatoid arthritis, psoriasis, treated autoimmune thyroiditis, or controlled Type 1 diabetes are acceptable)
6. History of human immunodeficiency virus (HIV), hepatitis B, or any active infection during Screening
7. History of cancer within 5 years of Screening, with the exception of fully treated non-melanoma skin cancers
8. Receipt of an experimental agent within 30 days or 5 half-lives prior to Screening, whichever is longer
9. Prior treatment with an immunomodulator other than a JAK inhibitor within 6 months of Screening; patients taking JAK inhibitors for AGS must have been on a stable dose for one month prior to Screening
10. Current treatment with a nucleoside reverse transcriptase inhibitor (NRTI) or other antiviral drug
11. Receipt of systemic corticosteroids within 30 days prior to Screening
12. Any vaccination within 30 days prior to Screening

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in innate immune signaling | 48 weeks
  Assessed by the expression of 30 interferon-stimulated genes (ISG), used to calculate an Interferon (IFN) score in whole blood
Incidence and severity of spontaneously reported treatment-emergent adverse events (TEAEs) of TPN-101 | 48 weeks
  Incidence and severity of spontaneously reported treatment-emergent adverse events (TEAEs) of TPN-101 administered for up to 48 weeks in patients with AGS

CONTACTS AND LOCATIONS:
Locations (5):
- Laboratory of Neurogenetics and Neuroinflammation Imagine Institute - INSERM U1163, Paris, France
- Italy (3):
  - Istituto Neurologico Casimiro Mondino, Pavia, Pavia
  - Presidio Ospedale dei Bambini [Children's Hospital], Brescia
  - SST Fatebenefratelli Sacco, Milan
- Royal Hospital for Children and Young People, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No